CLINICAL TRIAL: NCT04997005
Title: Prospective, Multicentre, Open Study Evaluating the Performance and Stability of the AMIStem-P Femoral Stem
Brief Title: The Medacta International AMIStem-P Post-Marketing Surveillance Study
Status: Active, not recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.001.16
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Arthrosis; Traumatic Arthritis; Rheumatoid Polyarthritis; Congenital Hip Dysplasia; Avascular Necrosis of the Femoral Head
MeSH Terms: conditions — Osteoarthritis; Hip Dislocation, Congenital; Femur Head Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: AMIStem-P — Performance of Total Hip Arthroplasty (THA) with AMIStem-P femoral stem implant

SUMMARY:
This is a Post-Market Surveillance study of AMIStem-P femoral stem prosthesis

ELIGIBILITY:
Inclusion Criteria:

* Patients with a disease (primary coxarthrosis, inflammatory arthritis of the hip, necrosis of the femoral head, etc.) requiring a total hip replacement
* Patient eligible to receive an uncemented AMIStem-P femoral stem
* Patient agreeing to comply with the study requirements
* Patient willing to provide written informed consent
* Patient affiliated to a social security system
* Patients between 18 and 85 years old

Exclusion Criteria:

* Participation in biomedical research
* Patients younger than 18 years old
* Vulnerable adult patients according to article L1121-6 of the French Public Health Code
* Pregnant or breastfeeding women
* Patients unable to provide written informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring Total Hip Arthroplasty and who are suitable to receive Medacta AMIStem-P femoral stem will be proposed to take part to the current post-market surveillance study during their pre-operative visit.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival rate | 10 years
  Kaplan Meier method

SECONDARY OUTCOMES:
Harris Hip Score | 3/6 months, 1, 3, 5 and 10 years
  Harris Hip Score [min = 0 (worst clinical outcome), max = 100 (best clinical outcome)]
Oxford Hip Score | 3/6 months, 1, 3, 5 and 10 years
  Oxford Hip Score [min = 0 (worst functional outcome), max = 48 (best functional outcome)]
Radiographic performance of the implants | 3/6 months, 1, 3, 5 and 10 years
  Presence of radiolucencies, migration, loosening, subsidence, tilt
Quality of life - Euroqol questionnaire | 3/6 months, 1, 3, 5 and 10 years
  EQ-5D-5L score [min = -0.59 (worst functional outcome), max = 1 (best functional outcome)]
Adverse events | intraop, 3/6 months, 1, 3, 5 and 10 years
  Intraoperative and postoperative adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Alexandru Nebunescu-Schirliu, MD, Principal Investigator — Hôpital Jacques-Puel
Locations (5):
- France (5):
  - Clinique de Saint Omer, Blendecques
  - Hôpital Castres, Castres
  - Nouvelle Clinique Bordeaux Tondu, Floirac
  - Clinique d'Orange, Orange
  - Hôpital Jacques-Puel, Rodez